CLINICAL TRIAL: NCT04663932
Title: Primary FIbrinolysis and Secondary STenting Versus immEdiate Stenting in ST-segment Elevation Myocardial Infarction (FISSTEMI)-- A Prospective Randomized Trial of Stent Implantation Strategy After Thrombolytic Therapy
Brief Title: Primary FIbrinolysis and Secondary STenting Versus immEdiate Stenting in ST-segment Elevation Myocardial Infarction
Acronym: FISSTEMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Collaborators: Tasly Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Yu Bo, The Second Affiliated Hospital of Harbin Medical University, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FISSTEMI-phase I
Record Dates: First submitted 2020-11-25; First posted 2020-12-11 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Acute Coronary Syndrome; Heart Diseases; Syndrome Heart Disease; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Coronary Disease; Vascular Diseases
Keywords: ST Elevation Myocardial Infarction; Microcirculatory dysfunction; Percutaneous coronary intervention; fibrinolysis
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Acute Coronary Syndrome; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Coronary Disease; Vascular Diseases; ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Eligible patients with STEMI who meet the Inclusion/Exclusion Criteria will receive thrombolytic therapy, and then be transferred to the PCI center for coronary angiography (CAG). Patients having a target vessel with TIMI grade 3 flow as shown by CAG, and and ≥ 50% angiographic stenosis after thrombus aspiration, will be randomized in a 1:1 ratio to either an immediate stenting group or a deferred stenting group. Patients assigned to the immediate stenting group will undergo appropriate stent implantation based on characteristics of the lesions. Patients assigned to the deferred stenting group will be sent back to the ward after PCI to receive standard anticoagulant and antiplatelet therapies, and the CAG will be repeated 5 to 7 days after initial intervention, followed by treatment with stent implantation.
Masking Description: This study is a prospective, multicenter, randomized, controlled, open-label clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate stenting group (Placebo Comparator): Patients assigned to the immediate stenting group will undergo appropriate stent implantation based on characteristics of the lesions.
  Interventions: Procedure: immediate stenting group(one-step strategy)
- deferred stenting group (Experimental): Patients assigned to the deferred stenting group will be sent back to the ward after PCI to receive standard anticoagulant and antiplatelet therapies, and the CAG will be repeated 5 to 7 days after initial intervention, followed by treatment with stent implantation.
  Interventions: Procedure: deferred stenting group (two-step strategy)

INTERVENTIONS:
Procedure: immediate stenting group(one-step strategy) — Patients assigned to the immediate stenting group will undergo appropriate stent implantation based on characteristics of the lesions.
  Other Names: Immediate Angioplasty
  Arms: immediate stenting group
Procedure: deferred stenting group (two-step strategy) — Patients assigned to the deferred stenting group will be sent back to the ward after PCI to receive standard anticoagulant and antiplatelet therapies, and the CAG will be repeated 5 to 7 days after initial intervention, followed by treatment with stent implantation.
  Other Names: Delayed angioplasty
  Arms: deferred stenting group

SUMMARY:
This prospective, multicenter, randomized, controlled, open-label clinical study has a target enrollment of 240 subjects. It will explore whether STEMI patients transferred to a PCI center following thrombolytic therapy and expected to have stent implantation might benefit from an alternative treatment strategy and the use of new technologies designed to improve myocardial protection throughout the medical care process.

DETAILED DESCRIPTION:
Eligible patients with STEMI who meet the Inclusion/Exclusion Criteria will receive thrombolytic therapy, and then be transferred to the PCI center for coronary angiography (CAG). Patients having a target vessel with TIMI grade 3 flow as shown by CAG, and and ≥ 50% angiographic stenosis after thrombus aspiration, will be randomized in a 1:1 ratio to either an immediate stenting group or a deferred stenting group. Patients assigned to the immediate stenting group will undergo appropriate stent implantation based on characteristics of the lesions. Patients assigned to the deferred stenting group will be sent back to the ward after PCI to receive standard anticoagulant and antiplatelet therapies, and the CAG will be repeated 5 to 7 days after initial intervention, followed by treatment with stent implantation.

All subjects will be recorded postoperative microcirculation perfusion and ST-segment drop of electrocardiogram and followed up by telephone or in the clinic at 1, 6, and 12 months after discharge from the hospital to obtain information including their general condition, chief complaints or discomforts, details of taking their oral medications, recent relevant test results, and to evaluate the primary endpoint, secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients who meet all of the following criteria can be included in the study:

  1. Age: 18-75 years old;
  2. A confirmed diagnosis of STEMI with symptom onset within 12 h;

STEMI criteria:

1. Patient has a history of chest pain/discomfort;
2. ST elevation ≥ 0.1 mV in at least two contiguous leads of an ECG on admission (> 30 minutes; ≥ 0.2 mV required for V2 and V3 ) or the development of new left bundle branch block (LBBB);
3. an increase in cardiac biomarkers (troponin, CK-MB) above the 99th percentile of the laboratory upper reference limit; 3. Time from FMC to wire crossing estimated to be > 120 min; 4. Has a target vessel with TIMI grade 3 flow shown as by CAG and ≥ 50% angiographic stenosis after thrombus aspiration; 5. Has culprit lesions identified as primary lesions; 6. Signed the written informed consent form.

Exclusion Criteria:

* Patients are not eligible for enrollment if they meet any of the following criteria:

  1. A contraindication to thrombolysis;
  2. An estimated survival time ≤ 12 months;
  3. Known heart failure of Killip class III or above, or mechanical complications such as heart rupture;
  4. Known to be participating in any other clinical trial;
  5. Pregnant or lactating women, or women experiencing their menstrual period;
  6. Weight < 40 Kg or > 125 Kg;
  7. Known allergies to drugs that are required during the study such as contrast agents, antiplatelet drugs, and anticoagulants;
  8. A target vessel with TIMI grade 0-2 flow as revealed by the initial CAG;
  9. Having lesions located in the LMCA or root of the LAD, or with severe multiple vessel disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Complete microvascular perfusion of subepicardial and myocardial tissues-TIMI flow grade 3 | one minute after the end of the each procedure
  Complete microvascular perfusion of subepicardial and myocardial tissues: TIMI flow grade 3 and TMP grade 3 and complete ST resolution on an ECG at 60 minutes after study intervention (STR ≥ 70%).
  For the immediate stenting group, the TIMI flow grade will be evaluated immediately after stent implantation. For the deferred stenting group, the TIMI flow grade will be evaluated after the first and second operations.
Complete microvascular perfusion of subepicardial and myocardial tissues-TMP grade 3 | one minute after the end of the each procedure
  Complete microvascular perfusion of subepicardial and myocardial tissues: TIMI flow grade 3 and TMP grade 3 and complete ST resolution on an ECG at 60 minutes after study intervention (STR ≥ 70%).
  For the immediate stenting group, the TMP grade will be evaluated immediately after stent implantation. For the deferred stenting group, the TMP grade will be evaluated after the first and second operations.
Complete microvascular perfusion of subepicardial and myocardial tissues-complete ST resolution on an ECG | within 60 minutes after PCI.
  Complete microvascular perfusion of subepicardial and myocardial tissues: TIMI flow grade 3 and TMP grade 3 and complete ST resolution on an ECG at 60 minutes after study intervention (STR ≥ 70%).
  All patients will have an 18-lead ECG within 60 minutes after PCI.

SECONDARY OUTCOMES:
TIMI flow grade for infarct-related arteries | one minute after the end of the each procedure
  For the immediate stenting group, the TIMI flow grade will be evaluated immediately after stent implantation. For the deferred stenting group, the TIMI flow grade will be evaluated after the first and second operations.
TIMI myocardial perfusion (TMP) grade for infarct-related arteries | one minute after the end of the each procedure
  For the immediate stenting group, the TMPG will be evaluated immediately after stent implantation. For the deferred stenting group, the TMPG will be evaluated after the first and second operations.
Measurement of ST resolution on an ECG | 60 minutes after PCI
  All patients will have an 18-lead ECG within 60 minutes after PCI.
TIMI myocardial blush grade (MBG) for infarct-related arteries | one minute after the end of the each procedure
  For the immediate stenting group, the MBG will be evaluated immediately after stent implantation. For the deferred stenting group, the MBG will be evaluated after the first and second operations.
Corrected TIMI frame count (cTFC) for infarct-related arteries | one minute after the end of the each procedure
  For the immediate stenting group, the cTFC will be evaluated immediately after stent implantation. For the deferred stenting group, the cTFC will be evaluated after the first and second operations.
TIMI myocardial perfusion frame count (TMPFC) | before and after each operation
  All subjects were required to calculate the preoperative and postoperative TMPFC (the delayed group was required to record the TMPFC before and after two operations respectively).
Myocardial infarct size | five to seven days after the last intervention (prior to discharge)
  The infarct area will be determined using semi-automatic contortion in the late short-axis enhanced image and will be expressed as a left ventricular mass percentage (%LV).
  2. Five to seven days after the first STEMI intervention (prior to discharge after delayed stent implantation), the myocardial infarct size will be recorded.
Myocardium salvage index (MSI) | five to seven days after the last intervention (prior to discharge)
  1. MSI refers to the ratio of rescue myocardium to AAR, which is a sensitive method to evaluate the effect of treatment.
  2. Five to seven days after the first STEMI intervention (prior to discharge after delayed stent implantation), the MSI will be recorded.

OTHER OUTCOMES:
All-cause death | 1, 6, and 12 months
  All deaths will be considered to be cardiac deaths unless a clear non-cardiac cause is identified.
  Patients will be followed up by telephone or in the clinic at 1, 6, and 12 months after discharge from the hospital to obtain information about all-cause death.
New or aggravated heart failure NYHA class IV | 1, 6, and 12 months
  Patients with cardiac disease that makes them unable to perform any physical activity without discomfort. Symptoms of heart failure may be present even at rest. If any physical activity is undertaken, discomfort is increased.
  Patients will be followed up by telephone or in the clinic at 1, 6, and 12 months after discharge from the hospital to obtain information about new or aggravated heart failure NYHA class IV.
Non-fatal re-infarction or revascularization of any acute infarct-related artery | 1, 6, and 12 months
  Myocardial infarction related to restenosis: angiographic restenosis ≥ 50% (complex lesions not found) after one stent implantation or balloon angioplasty procedure, accompanied by an elevation and/or decrease of cTn values in the absence of another occlusion.
  Patients will be followed up by telephone or in the clinic at 1, 6, and 12 months after discharge from the hospital to obtain information about non-fatal re-infarction or revascularization of any acute infarct-related artery.
Cardiogenic shock (1, 6, and 12 months after postoperation) | 1, 6, and 12 months
  Cardiogenic shock: systolic blood pressure < 90 mmHg, urine volume < 20 mL/h, clammy skin, cyanosis, tachypnea, and a pulse rate > 100 bpm.
  Patients will be followed up by telephone or in the clinic at 1, 6, and 12 months after discharge from the hospital to obtain information about cardiogenic shock.
Bleeding complications (classified as GUSTO) | 1, 6, and 12 months
  1. Severe or life-threatening: intracerebral hemorrhage or bleeding that results in substantial hemodynamic compromise requiring treatment;
  2. Moderate: bleeding that requires blood transfusion but does not result in hemodynamic compromise;
  3. Mild: bleeding that does not meet above criteria.
  4. Patients will be followed up by telephone or in the clinic at 1, 6, and 12 months after discharge from the hospital to obtain information about bleeding complications.
Stroke | 1, 6, and 12 months
  Stroke is defined as a sudden onset of focal neurological deficits due to cerebrovascular lesions, which lasts > 24 hours. Stroke is caused by ischemic or hemorrhagic cerebrovascular disorders.
  Patients will be followed up by telephone or in the clinic at 1, 6, and 12 months after discharge from the hospital to obtain information about stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided